CLINICAL TRIAL: NCT03986502
Title: Pilot Randomized Study of a Proactive Financial Navigation Intervention in Patients With Newly Diagnosed Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma
Brief Title: Financial Navigation Intervention in Improving Financial and Clinical Outcomes in Patients With Newly Diagnosed Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1005389; NCI-2019-03381 (Registry Identifier: NCI / CTRP); 10200 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-06-10; First posted 2019-06-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (financial navigation program) (Experimental): Patients and caregivers watch a web-based financial literacy video and receive information about financial counseling, direct medical cost and healthcare coverage assistance, and indirect and non-medical cost assistance.
  Interventions: Other: Media Intervention; Other: Informational Intervention; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Arm II (usual care) (Active Comparator): Patients and caregivers participate in usual clinic procedures and utilize any available clinic or community-based financial resources. Patients and caregivers will also be provided the financial navigation videos and worksheets from the intervention.
  Interventions: Other: Best Practice; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Media Intervention — Watch web-based financial literacy video
  Arms: Arm I (financial navigation program)
Other: Informational Intervention — Receive information on financial counseling and medical cost assistance
  Arms: Arm I (financial navigation program)
Other: Best Practice — Utilize usual clinic procedures and clinic or community-based financial resources
  Other Names: standard of care; standard therapy
  Arms: Arm II (usual care)
Other: Questionnaire Administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This trial studies how well a financial navigation intervention works in improving financial and clinical outcomes in patients with newly diagnosed gastric or gastroesophageal junction adenocarcinoma. Financial toxicity is a term used to summarize cancer-related financial hardship, including both the material (e.g. debt) and psychological (e.g. anxiety about costs) aspects. Cancer patients who experience financial toxicity are at greater risk for treatment non-adherence, poorer quality of life, and worse survival. Caregivers also share in this experience of financial toxicity and often spend money on food, medications, and other patient needs in addition to taking time off from work to provide logistical, emotional, and medical support. Financial navigation interventions that address the shared household financial concerns of patients and their caregivers may not only improve the patient outcomes but also improve caregiver burden, quality of life, and ability to perform caregiver roles more effectively.

DETAILED DESCRIPTION:
OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I (FINANCIAL NAVIGATION PROGRAM): Patients and caregivers watch a web-based financial literacy video and receive information about financial counseling, direct medical cost and healthcare coverage assistance, and indirect and non-medical cost assistance.

ARM II (USUAL CARE): Patients and caregivers participate in usual clinic procedures and utilize any available clinic or community-based financial resources.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT: English-speaking
* PATIENT: Diagnosis of gastric and/or gastroesophageal junction (GEJ) adenocarcinoma within 6 months of consent (any stage)
* PATIENT: Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* PATIENT: Receiving (or will receive) chemotherapy, radiation, or other systemic therapy (including targeted drug or immune checkpoint inhibitor)
* CAREGIVER: English-speaking

Exclusion Criteria:

• PATIENT: Enrolled in hospice care at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants that have experienced Household financial hardship | Up to 6 months
  Financial Hardship is defined as self-report of accrual of debt, taking out loans for cancer treatment or decline in household income <=20%
Patient quality of life: FACT-G | Baseline up to 6 months
  Composite score from the FACT-G. A 6-point score change is considered clinically meaningful in US cancer populations.
Subjective financial distress | Baseline up to 6 months
  Assessed using Comprehensive Score for Financial Toxicity-Patient Reported Outcome Measure (COST-FACIT). Mean scores (and standard deviations) at 3 and 6 months will be compared between intervention and control patients and caregivers using two sample t tests. Additionally, will explore the extent to which subjective financial distress correlates with financial hardship by comparing mean scores in those who experience financial hardship in each study arm versus those who do not.
Qualitative assessment of usual care and intervention | Up to 6 months
  Usual care arm dyads will be surveyed about availability (or lack), access to, and use of financial assistance via the clinic and community. Intervention arm dyads will be surveyed about availability and use of financial assistance from the clinic, community, and navigation partners. Will evaluate Consumer Education and Training Services (CENTS)'s and Patient Advocate Foundation (PAF)'s documentation and characterize the interventions made on behalf of dyads in subgroups categorized by age, gender, income, and financial fragility. We will review all unresolved issues reported by CENTS and PAF and describe the frequency and type by subgroup. We will describe dyads' use of clinic and community-based financial assistance resources in both study arms across subgroups, noting barriers to access if present.
Caregiver quality of life | Baseline up to 6 months
  City of Hope Quality of Life Family version, a well-validated tool with 37 items and 4 subscales (scored 0-10 per item). A change in score of 2 points per item is considered clinically meaningful.
Caregiver burden | Baseline up to 6 months
  Assessed via the social well-being subscale of the City of Hope Quality of Life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Veena Shankaran, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bell-Brown A, Hopkins T, Watabayashi K, Overstreet K, Leahy A, Bradshaw E, Gallagher K, Obenchain J, Padron A, Scott B, Flores B, Shankaran V. A proactive financial navigation intervention in patients with newly diagnosed gastric and gastroesophageal junction adenocarcinoma. Support Care Cancer. 2024 Feb 24;32(3):189. doi: 10.1007/s00520-024-08399-1. PMID 38400905

DOCUMENTS (1):
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03986502/ICF_000.pdf